CLINICAL TRIAL: NCT00540475
Title: The Pennsylvania Idiopathic Pulmonary Fibrosis State-wide Research Registry
Brief Title: Pennsylvania Idiopathic Pulmonary Fibrosis Research Registry
Acronym: PA-IPF
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Temple University (Other); University of Pennsylvania (Other); Geisinger Clinic (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kevin F. Gibson, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO07040328
Record Dates: First submitted 2007-10-03; First posted 2007-10-08 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Pennsylvania Idiopathic Pulmonary Fibrosis State-wide Research Registry (PA-IPF) is a cooperative project between five medical centers to coordinate a team of investigators. The aim of this registry will be: 1) To assess the extent of lung fibrosis in the commonwealth of Pennsylvania 2) To provide better access of patients with pulmonary fibrosis in all regions of Pennsylvania to standard of care and diagnosis 3) To facilitate the translation of new therapeutic interventions from the bench to the bedside.

DETAILED DESCRIPTION:
The University of Pittsburgh Medical Center, Dorothy P. & Richard P. Simmons Center for Interstitial Lung Disease is the coordination center for the Pennsylvania Idiopathic Pulmonary Fibrosis Statewide Research Registry, the collaborative institutions include: the University of Pennsylvania Health System, Geisinger Health System, and Penn State Milton S. Hershey Medical Center.

The PA-IPF Registry developed into a web site that contains information for patients, health professionals, and families, as well as an Internet-based database that will store information about patients to provide them with guidance about care, research, and support groups close to the area in which they live.

Benefits for membership in the PA-IPF Registry include:

* Staying informed about IPF research news, both nationally and locally.
* Having advance notice of any IPF research in which patients may be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis
* Sufficient testing results completed for an IPF Diagnosis (screening script)
* Adults (age > 18 years old)
* Participants who read and comprehend English language

Exclusion Criteria:

* Children
* Prisoner-patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2007-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
IPF Disease Course | 5 years
  Monitor IPF disease course

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — Medical Director, Dorothy P. & Richard P. Simmons Center
Locations (5):
- United States (5):
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Dorothy P. & Richard P. Simmons Center for Interstitial Lung Disease, Pittsburgh, Pennsylvania
  - The Center for Health Research at Giesinger Health System, Wilkes-Barre, Pennsylvania